CLINICAL TRIAL: NCT04709159
Title: Impact of Mobile Health Interactive Software on Tuberculosis Treatment Outcomes: The Call for Life (CFLU-TB) Project
Brief Title: Impact of Mobile Health Interactive Software on Tuberculosis Outcomes; The Call for Life (CFLU-TB) Project
Acronym: CFLU-TB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ST/263/2020
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Tuberculosis
Keywords: mHealth; Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis | interventions — CD56 Antigen

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with two arms. Interventional Arm will receive the intervention (daily pill reminders, health messages, clinic appointment reminders, remote symptom reporting service, toll-free number to call in to receive services, plus the option to co-register a caregiver who will receive the same services as the patient) as well as standard of care. The Control arm will have patients who will receive only standard of care available at the TB clinics as per the Uganda National Tuberculosis Treatment guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Participants on this arm will use Interactive Voice Response (IVR) daily pill reminders, thrice-weekly health messages, clinic appointment reminders, remote symptom reporting service and a 24 hour toll-free number to access services. These participants will also have the option to co-register a caregiver who will also receive daily pill reminders, clinic appointment reminder, weekly health tips and remote symptom reporting service.
  In addition, these participants will receive the standard of care according to Uganda National Tuberculosis Treatment guidelines.
  Interventions: Other: Call for Life Uganda
- Standard (No Intervention): These participants will receive the standard of care according to Uganda National Tuberculosis Treatment guidelines.

INTERVENTIONS:
Other: Call for Life Uganda — Call for Life™ Uganda (C4LU) is a web-based mHealth tool that provides treatment support to patients in the form of daily or weekly pill adherence reminders, health messages, clinic appointment reminders and a remote symptom reporting service. The tool interacts with patients by text message (SMS) or using voice and tone input via keypad (Interactive Voice Response - IVR) on both analogue and smart phones.
  The tool uses CONNECT FOR LIFE technology, which is on an open source platform developed by Grameen Foundation and the University of Southern Maine with financial support from the Bill and Melinda Gates Foundation. It was supported by Janssen, the Pharmaceutical Companies of Johnson and Johnson and was released under the terms of the MOTECH open source license agreement.
  Other Names: CONNECT FOR LIFE
  Arms: Intervention

SUMMARY:
This study will be an open-label Randomized Controlled Trial (RCT) to determine the effect of Call for Life TB (CFLU-TB) on Tuberculosis (TB) treatment success in patients with non-drug resistant Tuberculosis receiving care at three public health facilities, Kisenyi Health Centre IV, Kasangati Health Centre IV and Kiryandongo government Hospital.

Call for Life TB will employ a mobile health Health technology called CONNECT FOR LIFE™ to provide SMS or Interactive Voice Response patient support. This support will be in the form of clinic appointment, daily pill reminders, reminders, health tips and an opportunity to report symptoms which are responded to by a call from study doctors.

Collectively, 274 patients will be randomized (1:1ratio) to Intervention Arm (daily adherence calls, a pre-appointment reminder call, health tips and 24hr symptom reporting) or Standard of care (standard practice according to the national guidelines for TB treatment). Call for Life TB will also provide for Treatment supporters of patients on the Intervention Arm to be co-registered onto the system so as to enhance Directly Observed Treatment (DOTS).

Participants will be followed up for 6 months and observational data collected at several points. Data on sociodemographics, treatment response/outcome determined at 2 and at the end of treatment. Investigators shall conduct Focus Group Discussions (FGDs) and In- Depth Interviews (IDIs) with patients and clinic staff respectively, on ease of use, acceptability and satisfaction with the intervention.

Investigators will use system data to assess uptake and adherence to the tool. Investigators shall determine differences in the proportions of patients with treatment success in the two arms. Additionally, investigators shall assess adherence to medication, TB cure rates and treatment completion. Investigators shall qualitatively determine, perception, acceptability, and satisfaction with CFLU-TB. As a measure of cost-effectiveness, investigators shall determine marginal cost effectiveness CFLU-TB with regard to treatment success. The proposed study endpoint is 6-months retention in care, treatment and appointment adherence.

DETAILED DESCRIPTION:
Objectives of the study:

To determine the effect of CFLU-TB on TB treatment success (treatment completion and cure rates) in patients with TB receiving care at three public health facilities in Uganda.

Secondary Objectives

1. To compare TB cure rates (six months) in patients with microbiologically diagnosed TB.
2. To determine the effect of enhanced TB treatment support with CFLU-TB on 2- and 6-month retention in patients receiving TB treatment at Kisenyi Health Center IV.
3. To assess views of care-providers towards the CFLU-TB.
4. To assess the cost-effectiveness of the CFLU-TB intervention in TB care
5. To determine and compare adherence rates between patients in the intervention arm and control arms.
6. To compare treatment completion (six months) in patients clinically diagnosed with TB in the intervention and control arms.
7. To compare knowledge about TB/HIV in patients enrolled in the intervention and control arms.
8. To determine the effect of CFLU-TB on adherence to clinic appointments.
9. To determine the level of usage of the CFLU-TB tool in patients and their care providers
10. To determine rifampicin-resistance rates in the intervention and control arms.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of TB diagnosis-either confirmed bacteriologically by Xpert MTB/RIF Version G4 assay (Cepheid, Sunnyvale, CA, USA) or clinically diagnosed by health worker.
* Evidence of a personally signed and dated informed consent document indicating that the participant (or a legal representative) has been informed of all pertinent aspects of the study.
* Willingness to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Aged 18 years or more
* Mobile phone ownership
* Patients who can understand Luganda, Runyankole, Swahili or English. These languages are the languages spoken by of the majority of patients at three health. Other languages may be added to the service if the anticipated demand surpasses 30 patients.

Exclusion Criteria:

* Patient unable to use a basic feature phone or who whose clinical condition that interferes with appropriate use of cell phone for voice calls (e.g., deafness, severe cognitive impairment)
* Ongoing participation in another interventional study that the investigator believes will interfere with study procedures or assessment of outcomes of this study.
* Patients who are critically ill.
* Patients with drug resistant TB (Rifampicin resistant, Multi-drug resistant and Extensive drug resistant TB).
* Patients with TB Meningitis or Osteoarticular TB.
* Any other clinical condition that, in the opinion of the site investigator, would make the participant unsuitable for the study or unable to meet with dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Treatment success | After 6 months of treatment
  Percentage of patients with treatment success. Treatment success is the sum of the percentages of patients declared cured and those who complete treatment.

SECONDARY OUTCOMES:
TB cure for patients with bacteriologically diagnosed TB | After 6 months of treatment
  Percentage of cured patients. TB cure is a pulmonary TB patient with bacteriologically confirmed TB at the beginning of treatment who was smear- or culture-negative in the last month of treatment and on at least one previous occasion.
Treatment completion for patients with clinically diagnosed TB | After 6 months of treatment
  Percentage of patients who complete treatment.Treatment completion is a TB patient who completed treatment without evidence of failure BUT with no record to show that sputum smear or culture results in the last month of treatment and on at least one previous occasion were negative, either because tests were not done or because results are unavailable.
Retention in care | At 2 and 6 months
  Percentage of patients active in care. Retention in care is evidence of a clinic visit within 30 days of last visit appointment.
Experiences of patients and care providers towards CFLU™ | At baseline, 2 months and 6 months
  Themes discussed through Focus Group Discussions and In-Depth Interviews
Cost effectiveness of the CFLU™ intervention | At 6 months
  Incremental cost per additional DALY averted as a result of improvement in treatment success using governmental and societal perspective
Adherence to TB medicines | At 2 months and 6 months
  Mean adherence rates (proportion of TB medicines taken as evidenced by TB card
Appointment keeping | At 2 months and 6 months
  Proportions of patients who keep their appointment; proportions of early, on-time and late appointments)
Knowledge about HIV/TB | Continuous variable
  Mean increase in knowledge about TB/HIV
Drug resistant TB rates | At 5 months and 6 months
  Absolute numbers and proportions of patients with Rifampicin resistance by GeneXpert
Uptake of intervention | At 2 months, 4 months and 6 months
  Mean call success rate

CONTACTS AND LOCATIONS:
Overall Officials: Dathan Byonanebye Mirembe, MBChB, M.MED, Principal Investigator — Infectious Diseases Institute
Locations (3):
- Uganda (3):
  - Kasangati Health Centre IV, Kampala
  - Kisenyi Health Centre IV, Kampala
  - Kiryandongo Hospital, Kiryandongo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byonanebye DM, Mackline H, Sekaggya-Wiltshire C, Kiragga AN, Lamorde M, Oseku E, King R, Parkes-Ratanshi R. Impact of a mobile phone-based interactive voice response software on tuberculosis treatment outcomes in Uganda (CFL-TB): a protocol for a randomized controlled trial. Trials. 2021 Jun 13;22(1):391. doi: 10.1186/s13063-021-05352-z. PMID 34120649